CLINICAL TRIAL: NCT04644731
Title: ULTRA-Peds: A Multicenter Data Registry for Outcomes for Pediatric Volume Overload
Brief Title: Ultrafiltration Therapy Registry Using Aquadex (ULTRA-Peds)
Acronym: ULTRA-Peds
Status: Terminated | Type: Observational
Why Stopped: The study was stopped early only due to a business decision to pursue development of a pediatric dedicated device. This decision was not based on any efficacy or safety concerns."
Sponsor: Nuwellis, Inc. (Industry)
Collaborators: AKI Critical Care Research Foundation (Other)
Responsible Party: Sponsor
Other Study IDs: CLIN07423
Record Dates: First submitted 2020-11-10; First posted 2020-11-25 (Actual); Last update posted 2024-02-20 (Actual); Status verified 2024-02

CONDITIONS: Fluid Overload
MeSH Terms: conditions — Edema

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 90 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (1):
- Pediatric patients who require fluid removal: Pediatric patients who require fluid removal with the Aquadex™ System per local standard of care
  Interventions: Device: Aquadex™ System

INTERVENTIONS:
Device: Aquadex™ System — Ultrafiltration for fluid removal

SUMMARY:
The ULTRA-Peds registry will employ a multi-center, single-arm, open-label, observational design to capture baseline, procedural and follow-up data on pediatric patients that have been treated (i.e., retrospective data from treatment at the time of registry approval by the IRB) or are scheduled to be treated (i.e., prospective data for on-label treatment after registry approval by the IRB) with Aquadex therapy according to local standard of care practices and decisions. All prospective data will be from on-label Aquadex treatment of pediatric patients weighing 20 kilograms or more. No data from prospective off-label treatment (i.e., Aquadex treatment with other adjunctive or conjunctive therapies for pediatric patients who may weigh less than 20kg) will be included in the registry. An estimated 10 sites in the United States who have received training in extracorporeal therapy and the Aquadex™ system will enroll a minimum of 500 patients.

DETAILED DESCRIPTION:
The ULTRA-PEDs registry is designed to capture data in the real-World clinical setting on the Aquadex™ system in local standard of care, with the aim of understanding it's performance and utilization. Enrollment is expected to take approximately 2.5 years from the time the first patient is enrolled to the time the final patient is discharged from the hospital.

ULTRA-PEDs will allow prospective and retrospective data collection for the following scenarios:

* All prospective data for on-label use only (i.e., Aquadex ultrafiltration therapy for pediatric patients weighing 20 kg or more, whose fluid overload is unresponsive to medical management, including diuretics).
* Retrospective patients at the time of registry approval by IRB regardless of on-label or off-label use.

  * Retrospective on-label use
  * Retrospective off-label use (i.e., Aquadex ultrafiltration with other adjunctive or conjunctive therapies for pediatric patients who may weigh less than 20kg)

ELIGIBILITY:
Inclusion Criteria:

I. For enrollment in prospective data collection:

1. Patient age is 21 years or younger
2. Patient weighs 20 kilograms or more.
3. Patient or legally authorized representative provides written authorization or patient is hospitalized and receiving treatment in a center with an Institutional Review Board that has allowed for waived consent based on the type of data being collected for the Registry.
4. Patient is to undergo Aquadex therapy for fluid overload (i.e., fluid removal) as local standard of care.

II. For enrollment in retrospective data collection:

1. Patient age is 21 years or younger.
2. Patient or legally authorized representative provides written authorization or patient is hospitalized and receiving treatment in a center with an Institutional Review Board that has allowed for waived consent based on the type of data being collected for the Registry.
3. Patient underwent Aquadex therapy for fluid overload (i.e., fluid removal) as local standard of care.

Exclusion Criteria:

1. Unable or unwilling to provide informed consent
2. Unable or unwilling to comply with study requirements

Max Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Pediatric patients who require fluid removal with the Aquadex™ System per local standard of care
Sampling Method: Non-Probability Sample
Enrollment: 97 (Actual)
Dates: Start 2021-04-09 (Actual); Primary Completion 2023-09-13 (Actual); Study Completion 2023-09-13 (Actual)

PRIMARY OUTCOMES:
Treatment Survival | Through completion of a treatment course, up to 3 months
  Patient survive treatment course
Survival at ICU discharge | Through completion of a treatment course in the ICU, up to 1 month
  % of ICU patients survive treatment in ICU
Change in Kidney Function | Change eGFR and renal labs from initiation to completion of treatment, up to 3 months
  Assessment of Kidney function
Hemodynamic stability at initiation of UF therapy | From the time of index procedure is initiated up to 60 minutes after initiation
  Need resuscitation fluids and medications (e.g. vasoactive medication)
Hemodynamic stability during treatment course | Through completion of a treatment course, up to 3 months
  Need for vasoactive medication
Change % fluid overload during treatment course | Through completion of a treatment course, up to 3 months
  % change in weight from initiation to the end of the last Aquadex procedure
Length of Stay in ICU | The time from admission to ICU through discharge from ICU, usually 1 month
  Time of admission to ICU to discharge
Change in PRISM III Score | 2 hours before ICU admission through the first 4 hours after ICU discharge
  Physiologic variables and labs to assess mortality risk
Aquadex related adverse events | Through completion of a treatment course, up to 3 months
  Aquadex related adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Stuart Goldstein, MD, Study Chair — AKI Critical Care Research Foundation
Locations (7):
- United States (7):
  - Children's of Alabama Hospital, Birmingham, Alabama
  - Lucile Packard Children's Hospital Stanford, Palo Alto, California
  - Joe DiMaggio Children's Hospital, Hollywood, Florida
  - Riley Children's Hospital, Indianapolis, Indiana
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Le Bonheur Children's Hospital, Memphis, Tennessee
  - Seattle Children's Hospital, Seattle, Washington

IPD SHARING:
Plan to Share IPD: Undecided